CLINICAL TRIAL: NCT00615225
Title: Observational Study on the Systemic Inflammatory Response During Brain Death.
Brief Title: Brain Death: Inflammatory Response, Apoptosis, and Endotoxin Tolerance
Status: Completed | Type: Observational
Sponsor: Delafontaine Hospital (Other)
Responsible Party: Christophe Adrie, Delafotaine Hospital
Other Study IDs: CCPPRB/114-02; Agence de Biomédecine 2005
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-02

CONDITIONS: Brain Death
Keywords: brain death; inflammation; endotoxin; transplantation; graft; apoptosis; Systemic inflammatory response; Apoptosis activation; Graft outcome
MeSH Terms: conditions — Brain Death; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Brain dead patients: All patients meeting criteria for brain death
  Interventions: Procedure: Muscle biopsy
- Healthy control: Any healthy volunteers accepting to give some blood
- Volunteers having hip surgery: Patients undergoing hip surgery for degenerative non-inflammatory hip disease
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — Muscle biopsies were taken through the operation site from the vastus lateralis thigh muscle at the beginning of surgery
  Groups: Brain dead patients; Volunteers having hip surgery

SUMMARY:
We hypothesized that brain death is associated with an early systemic inflammatory response, possibly combined with activation of apoptotic cell death, two events that may contribute to induce rapid organ dysfunction. In this study of brain-dead donors and controls, we assayed plasma cytokines and soluble factors, investigated plasma endotoxin levels as a triggering factor for inflammation, measured ex vivo cytokine production by blood leukocytes to determine whether immunosuppression occurred after brain death, and examined skeletal muscle biopsies to look for evidence of inflammation and increased apoptosis in peripheral tissue.

ELIGIBILITY:
Inclusion Criteria:

* All brain dead patients whatever the cause (cardiac arrest, stroke, head trauma)

Exclusion Criteria:

* Age < 18years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any brain dead patients diagnosed in three different ICUs
Sampling Method: Non-Probability Sample
Dates: Start 2000-01; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Adrie, MD, PhD, Principal Investigator — Delafontaine Hospital; Jean Marc Cavaillon, ScD, Study Director — Pasteur Institute
Locations (3):
- Liege Hospital, Liège, Belgium
- France (2):
  - Tenon Hospital, Paris
  - Delafontaine Hospital, Saint-Denis